CLINICAL TRIAL: NCT00523471
Title: Gamma-H2AX as a Molecular Predictor of Prostate Cancer Radiosensitivity
Brief Title: Blood Test to Measure DNA Damage in Blood
Status: Terminated | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: GU-6-0076/ethics 23586
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; gamma H2AX; radiosensitivity
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood test

SUMMARY:
To check the radiosensitivity level in individual patients based on their DNA damage level.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer diagnosis
* undergoing radiotherapy
* agree to participate in study

Exclusion Criteria:

* not willing to participate
* not undergoing radiotherapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Pervez, MBBS, FRCPC, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada